CLINICAL TRIAL: NCT05236049
Title: Evaluation of Safety and Efficacy of Wrapping Orbital Implant by SclerFIX Product After Eye Enucleation
Brief Title: Use of an Allograft Set-up (SclerFIX) as Replacement of Sclera Graft for Support of Enucleation Implant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SclerFIX-TBF1; 2018-A01738-47 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-01-03; First posted 2022-02-11 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Enucleated; Eye; Eye Cancer
MeSH Terms: conditions — Eye Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SclerFIX (Experimental): Strip of umbilical cord lining membrane allograft wrapped around the bioceramic enucleation implant. The assembly is placed inside the void orbital cavity and the muscles are sutured to the SclerFIX strips.
  Interventions: Biological: SclerFIX

INTERVENTIONS:
Biological: SclerFIX — Chemically-treated, viro-inactivated, freeze-dried and irradiated umbilical cord lining membrane allograft used as substitute for scleral graft in support of intraocular implant.

SUMMARY:
The purpose of this open, monocenter pilot trial is to evaluate the tolerance of the SclerFIX product, an allograft of umbilical cord lining membrane, in the reinforcement of ocular implants in patients who underwent enucleation due to an eye malignant tumor resection.

DETAILED DESCRIPTION:
As scleral graft is forbidden in France, it cannot be used for support of enucleation implants. This study investigational product, SclerFIX, was developed to substitute scleral grafts in those cases.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 45 and 85 years old, presenting an enucleation caused by malignant tumor resection.
* Oncological treatment compatibility with enucleation and intra-orbital implant.
* Surgery requiring the placement of an enucleation implant.
* Persistence of the oculomotor muscles allowing their insertion into the tissue.
* Patient with social security coverage.
* Consenting and informed patient.

Exclusion Criteria:

* Pregnant or breast-feeding women: women of childbearing age were asked to undergo a pregnancy test before being enrolled into the study and to use an effective birth control method.
* Patient presenting an infectious risk (neutropenia, active local infection, immunodeficiency).
* Patient with autoimmune disease.
* Proton-therapy / radiotherapy of the eye before healing.
* Patient with oculomotor muscles invasion or non-attachment of these muscles.
* Allergy to contrast agents used in radiology.
* Patient under legal guardianship.
* Patient not benefiting from the social security cover.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Number of complications and adverse events related to SclerFIX set-up as replacement of sclera graft for support of enucleation implant | Through study completion (6 months)
  Evaluation of SclerFIX tolerance by physical examination of the patient: clean scar; absence of redness, edema, ulcer, granuloma and cystic lesion; absence of signs of protrusion and inflammation

SECONDARY OUTCOMES:
Rate of integration of SclerFIX set-up in the orbital cavity with muscles attachment allowing enucleation implant mobility | 7 days, 15 days, 1 month, 3 months, 6 months
  Evaluation by physical examination by the surgeon of the set-up assembly and its maintenance over time with insertion of oculomotor muscles, integration of these latter, and maintenance of the movement of the implant
Evaluation of surgical wrapping and attachment with muscles | Time of investigational product surgical implantation (Day 0)
  Surgeon assessment on completeness and difficulty of oculomotor muscles insertion at the time of product implantation (Day 0)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: No